CLINICAL TRIAL: NCT02164058
Title: A Randomized Controlled Multicenter Study on the Use of the TandemHeart to Reduce Infarct Size
Brief Title: TandemHeart to Reduce Infarct Size (TRIS Trial)
Acronym: TRIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: CardiacAssist, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA 2011-01
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial infarction; STEMI; ST elevation MI; Acute MI
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TandemHeart System + PCI (Experimental): TandemHeart System prior to percutaneous coronary intervention
  Interventions: Device: TandemHeart System; Procedure: Percutaneous coronary intervention
- PCI (Active Comparator): Percutaneous coronary intervention
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Device: TandemHeart System
  Arms: TandemHeart System + PCI
Procedure: Percutaneous coronary intervention
  Other Names: PCI

SUMMARY:
The purpose of this study is to determine if a device known as the TandemHeart® System (TandemHeart) can help limit heart damage and reduce serious complications after a certain type of heart attack (acute ST elevation anterior wall myocardial infarction [STEMI]) by evaluating the use of the TandemHeart system prior to a procedure called percutaneous coronary intervention (PCI)

ELIGIBILITY:
INCLUSION CRITERIA

The following is a list of general inclusion criteria. More detailed information can be found in the study protocol.

1. ≥ 18 years of age
2. Presents within 6 hours of acute MI symptoms
3. Evidence of ST elevation
4. First myocardial infarction
5. Written informed consent

EXCLUSION CRITERIA

The following is a list of general exclusion criteria. More detailed information can be found in the study protocol.

1. Contraindications to antiplatelet/anticoagulation therapy
2. History of blood disorders or active bleeding
3. Renal dysfunction or failure
4. Neurologic damage
5. Cardiogenic shock
6. History of cerebrovascular disease
7. History of transfusion reaction
8. Prior coronary artery bypass surgery
9. Participation in another trial with an investigational drug or device
10. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | 30 days post-procedure
  Major Adverse Cardiac or Cerebrovascular Events (MACCE):
  * Death, all cause
  * Stroke
  * Reinfarction
  * Major vascular complications